CLINICAL TRIAL: NCT06760663
Title: The Load-velocity Relationship: Neuromuscular Adaptations to Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Afonso Fitas, Master of Science, University of Lisbon
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CEIFMH Nº 28/2023; 2023.02063.BD (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2024-10-05; First posted 2025-01-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Muscle Hypertrophy
Keywords: load-velocity relationship; neuromuscular; hypertrophy; strength; velocity-based training
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Intervention Model Description: Each of the 3 groups will perform 10 weeks of training. After all data is collected, it will be processed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Percentage Based-Training (PBT) (Active Comparator): Training load will be prescribed in a traditional fashion. No adjustments of load will be performed.
  Interventions: Behavioral: The load-velocity relationship: Neuromuscular adaptations to resistance training
- Velocity Based Training (VBT) (Experimental): Training load will be adjusted according to daily fluctuations in movement velocity.
  Interventions: Behavioral: The load-velocity relationship: Neuromuscular adaptations to resistance training
- Fast Velocity Based Training (VBT-F) (Experimental): Training load will be adjusted according to fluctuations in movement velocity. Repetitions will be performed as fast as possible.
  Interventions: Behavioral: The load-velocity relationship: Neuromuscular adaptations to resistance training

INTERVENTIONS:
Behavioral: The load-velocity relationship: Neuromuscular adaptations to resistance training — Comparing the impact of adjusting training load based on movement velocity on hypertrophy and neural adaptations.

SUMMARY:
Adaptations to resistance training are highly specific and depend on the combination of external loading and the level of individual adaptability. As the relationship between load and velocity of movement is strong and linear, the application of velocity-based training (VBT) has been proposed to enable load adjustments to ensure that exercise is performed at a given intensity independently of several factors such as fatigue. It was recently shown that VBT potentiates increases in muscle strength and power when compared to that seen following a percent-based training (PBT). As the development of muscle strength is explained by the combination of hypertrophy and heightened neural drive, it is important to unravel whether VBT is superior to PBT in eliciting positive adaptations at both these levels or exclusively at one of them. Thus, the aim of this study is to thoroughly compare the neuromuscular adaptations of VBT with the ones found in PBT.

DETAILED DESCRIPTION:
The primary aim of this project is to compare the effect of VBT with that of PBT on muscular hypertrophy and neuromuscular RT adaptations during an intervention of similar volume lasting 10 weeks. As a secondary purpose, the investigators also intend to examine the relationship between these adaptations with post-training gains in different forms of muscle strength (slow and fast-speed strength, as well as endurance muscle strength). As a tertiary purpose, the investigators aim at determining how neuromuscular fatigue, training stress and muscular damage evolve in response to VBT and PBT during the 10-week intervention. As a quaternary purpose, the investigators intend to assess if the results are consistent for both upper-body and lower-body RT exercises.

The investigators hypothesize that, after 10 weeks of RT, (i) despite showing larger increases in strength, power and muscular activation [increases in motor unit firing rate and recruitment due to high speed contractions ] , due to a lower level of mechanical tension during training , participants assigned to VBT will display less muscular hypertrophy; (ii) participants assigned to VBT will present larger increases in slow- and fast-speed strength and athletes assigned to PBT will present larger increases in endurance strength ; (iii) participants assigned to VBT will present less neuromuscular fatigue, training stress and muscular damage; (iv) the aforementioned hypothesized outcomes will be consistent for both upper- and lower-body RT exercises.

Research Plan and Methods Participants Recruitment Healthy male participants aged 18-30 years without neurologic conditions, lower and upper limb disabilities, or any known disease will be recruited. All participants must be familiar with RT (≥ 3 times per week, for at least 3 years of practice). Additional exclusion criteria will be known metabolic, cardiovascular, respiratory disorders or other orthopedic conditions that limit exercise. The participants will need to sign an informed consent before participation, already approved by the institutional review board (CEFMH Nº 28/2023).

Study Design Participants will be randomly allocated to one of three groups: PBT, VBT or VBT performed as fast as possible (VBT-F). All groups will entail a RT intervention and all groups will be assessed at baseline, 4 weeks, and 10 weeks (T0, T4, and T10, respectively).

Sample Size Justification Based on the effect size of the differences in the back-squat one-repetition maximum (1RM) after 6 weeks of PBT and VBT (and accounting for a 25% attrition rate due to the study's longitudinal nature) a total of 30 participants (10 per group) will be recruited to provide 95% statistical power .

RT Protocols RT will be performed 3 times per week, with a minimum of 48h rest between each session. Participants will perform 3 sets of repetitions of the free-weight back squat and free-weight bench press per session, with the number of sets incrementing by one each 2 weeks. , at a load corresponding to 85%1RM. VBT-F participants will perform the same number of sets and repetitions as those enrolled in PBT and VBT, with the concentric phase performed at maximal intended velocity. In both exercises, the eccentric phase will be performed in a non-explosive and controlled condition and without imposing a pause before the beginning of the concentric contraction. Exercise load will correspond to 85%, 77.5% and 70% of the 1RM on the first, second and third sessions of the week, respectively. The VBT and VBT-F group will adjust loads each session according to meaningfull fluctuations in MCV (0.06 m/s and 0.02 m/s for the squat and bench press, respectively). MCV will be monitored using a validated linear position transducer sampling the bar's velocity at a frequency of 1,000 Hz (Chronojump, Barcelona, Spain). Velocity feedback will be given to participants during RT sessions.

Testing

Testing will involve two sessions to avoid prolonged data collection and minimize mental and physical fatigue. Objective measures of strength, muscular and neurophysiological properties will be collected as briefly described below:

Muscle Hypertrophy Assessments of muscle cross-sectional area, muscle thickness, fascicle length and pennation angle will be conducted via ultrasonography [B-mode device (Noblus; Hitachi Aloka Medical Systems, Tokyo, Japan) with a linear-array probe (4.0 cm)] . Participants will be instructed to lie supine and relaxed. As the magnitude of muscle hypertrophy may differ between proximal and distal portions of the muscle, measurements will be performed at various sites of the quadriceps femoris and the pectoralis major.

Strength and Muscular Activation Back squat and bench press maximum voluntary isometric contractions (MVIC) will be conducted on a Smith-Machine (Matrix Fitness; G1 Smith machine, Cottage Grove, WI) coupled to a force plate with a sampling rate of 1,000 Hz (Bertec, Colombia, USA). Three MVICs will be performed, lasting 5 s each with a 60 s interval of rest between trials. Participants will be instructed to exert their maximum force as fast and hard as possible. Rate of force development will be calculated sequentially as the slope of force-time relationship during each MVIC trial (0-50, 50-100 and 100-150 ms after force onset). Then, a countermovement jump (CMJ) and a bench press-throw test, comprised of 3 attempts, will be performed to assess fast-speed strength. Additionally, 1RM will also be determined for the free-weight back squat and the free-weight bench press to assess slow-speed strength. 1RM will also be used to set the initial loads of the PBT intervention. 1RM will be defined as the maximal load mobilized throughout full range of motion in a single repetition. Lastly, participants will perform a set to volitional failure with a load corresponding to 60% 1RM for the back squat and bench press (endurance strength). Strong verbal encouragement will be provided for motivation. Surface electromyography (EMG) of the quadriceps femoris and pectoralis major will be used to quantify muscle activation during all testing sessions through bipolar wireless sensors (EMG Delsys, TrignoTM), sampled at a 1,000 Hz. Raw EMG data will be stored in digital format using the Acqknowledge 4.3.1 software (BIOPAC Systems Inc., Goleta, CA) and smoothed by root mean square (RMS) calculation. The RMS will be indicative of the amplitude of muscular activation and the RMS obtained in response to dynamic assessments will be normalized to that obtained at MVIC.

Training Stress, Neuromuscular Fatigue and Muscular Damage Each week, all participants will complete three CMJ. Additionally, participants will provide their rate of perceived exertion (RPE), on an increasing scale from 1-10, of each performed set during the RT intervention. Lastly, weekly assessments of capillary creatine kinase (CKMM) will be conducted. To determine CKMM activity, a sample of 32 μl of capillary blood will be collected from the ear lobe into a tube containing heparin (Cat n ° 9550532 Reflotron ®. These three assessments will be the indicators of neuromuscular fatigue, training stress and muscular damage, respectively, throughout the intervention .

Statistical Analysis All data will be presented as means and standard deviation and will be tested for normality and homoscedasticity with the Shapiro-Wilk and Levene's test, respectively. A two-way repeated measures ANOVA [condition (PBT vs. VBT-F vs. VBT) x time (T0 vs. T4 vs. T10)] will be used to explore main effects and interactions for each dependent variable. Adjustment of multiple comparisons will be made with Bonferroni's correction. Data analyses will be performed using SPSS software version 27.0 (SPSS Inc., Chicago, IL, USA) and statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without neurologic conditions;
* Individuals without lower and upper limb disabilities;
* Individuals without any known disease.;
* All participants must be familiar with Resistance Training (≥ 3 times per week, for at least 3 years of practice).

Exclusion Criteria:

* Individuals with known metabolic disease;
* Individuals with known cardiovascular disease;
* Individuals with respiratory disorders or other orthopedic conditions that limit exercise.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Pectoralis major cross sectional area | 10 weeks
  Measurements of cross sectional area of the right pectoralis major muscle
Quadriceps femoris cross sectional area | 10 weeks
  Cross sectional area of the right quadriceps femoris muscle
Quadriceps femoris muscular thickness | 10 weeks
  Muscular thickness f the right quadriceps femoris muscle
Pectoralis major muscular thickness | 10 weeks
  Muscular thickness of the right pectoralis major muscle

SECONDARY OUTCOMES:
Back Squat Maximal Strength | 10 weeks
  Measurement of maximal voluntary isometric contraction of the smith machine back squat
Muscular activation | 10 weeks
  Measurements of surface electromyography on the pectoralis major and vastus lateralis.
Bench Press Maximal Strenght | 10 weeks
  Measurement of the maximum voluntary isometric contraction of the smith machine bench
Back squat and bench press one-repetition maximum | 10 weeks
  Incremental loading protocol of the back squat and bench press exercises.
Back Squat and Bench Press Load-Velocity relationships | 10 weeks
  Measurement of the velocity at which different relative loads are lifted in the bench press and back squat exercises
Back squat and bench press strength endurance | 10 weeks
  Determination of the maximum number of repetitions performed at 60% of the one-repetition maximum of the bench press and back squat exercises
Countermovement jump height | 10 weeks
  Determination of the maximal achieved height of 3 attempts of the countermovement jump
Bench press throw height | 10 weeks
  Determination of the maximum height at which a weighted barbell can be thrown with 30, 40 and 50% of the one repetition maximum of the bench press

CONTACTS AND LOCATIONS:
Overall Officials: Gonçalo Mendonca, PhD, Study Director — Faculdade de Motricidade Humana - Universidade de Lisboa
Locations (1):
- Faculdade de Motricidade Humana Universidade de Lisboa, Cruz Quebrada, Oeiras, Portugal

IPD SHARING:
Plan to Share IPD: No